CLINICAL TRIAL: NCT03303196
Title: Bihormonal Bionic Pancreas for the Treatment of Diabetes Post-Pancreatectomy in Children With Congenital Hyperinsulinism - A Pilot Study
Brief Title: Bionic Pancreas in Children With Hyperinsulinism and Post-Pancreatectomy Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Boston University (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diva De Leon, MD, MSCE, Director, Congenital Hyperinsulinism Center, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-014144
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Hyperinsulinism; Diabetes; Pancreatic Diseases; Pancreatectomy; Hyperglycemia
Keywords: Post-Pancreatectomy Diabetes; Insulin Therapy
MeSH Terms: conditions — Hyperinsulinism; Diabetes Mellitus; Pancreatic Diseases; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: This will be an open-label, pilot clinical trial to assess efficacy and safety of the bihormonal bionic pancreas in children and young adults with HI who have developed post-pancreatectomy diabetes. Subjects will be studied during two research inpatient admissions at the CHOP HI Center. The order of the interventions will be randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Bihormonal bionic pancreas admission (Experimental): Four day inpatient admission where participants will have blood sugar managed by the Bihormonal Bionic Pancreas. Blood sugars will be monitored for safety by study staff.
  Interventions: Device: Bihormonal Bionic Pancreas
- Standard care admission (No Intervention): Four day inpatient admission where participants will have blood sugar managed by the participant's home-glucose control regimen. Blood sugars will be monitored for safety by study staff.

INTERVENTIONS:
Device: Bihormonal Bionic Pancreas — A 4-day inpatient admission in which subjects will wear the bihormonal pancreas. The bihormonal pancreas will be placed upon admission and there will be 1 day of run-in. This will be followed by 3 days of data collection for comparison with the data obtained from the standard of care during the control admission.
  Arms: Bihormonal bionic pancreas admission

SUMMARY:
This is a pilot study designed to determine if the bihormonal bionic pancreas provides improved blood glucose control, compared to the current standard of care, in individuals with hyperinsulinism who developed diabetes after having a pancreatectomy.

DETAILED DESCRIPTION:
The management of diabetes following pancreatectomy for hyperinsulinism (HI) generally consists of the same approaches that are used for individuals with type 1 diabetes (T1D). However, there are significant differences in individuals with HI and post-pancreatectomy diabetes that increases the risk of hypoglycemia in these individuals and prevent achieving tight glycemic control. Individuals with HI have glucagon deficiency and unlike T1D, those with HI and post-pancreatectomy diabetes have residual dysregulated insulin secretion that results in marked hypo- and hyper-glycemia. Furthermore, pancreatic insufficiency can result in disturbances in nutrient absorption and fluctuations in glucose concentrations.

Current treatment approaches with intermittent subcutaneous insulin administration or insulin pump therapy offer inadequate glycemic control in these individuals. We propose a novel approach to the management of these individuals with the bihormonal bionic pancreas to replace both hormones, insulin and glucagon, through an automated glycemic management system.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 6 to 30 years.
2. Diagnosis of hyperinsulinism.
3. Previous pancreatectomy.
4. Diabetes confirmed by one or more of the following:

   * Glycosylated A1c > 6.4%.
   * Fasting glucose > 125 mg/dL.
   * 2-hour post-prandial glucose > 200 mg/dL.
   * Random glucose > 200 mg/dL with symptomatic hyperglycemia.
5. On insulin therapy with a regimen of at least 11 units/kg/day.
6. Treatment with subcutaneous insulin by pump at the time of recruitment.
7. Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the site PI).
8. Females > 11 years of age must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
9. Informed consent, parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Unable to provide informed consent (e.g. impaired cognition or judgment).
2. Evidence of a medical condition that might alter results or compromise the interpretation of results, including active infection, kidney failure, severe liver dysfunction, severe respiratory or cardiac failure.
3. Evidence of severe hematologic abnormality including severe anemia and/or thrombocytopenia.
4. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to radio frequency interference.
5. Unable to completely avoid acetaminophen for duration of study.
6. History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
7. Established history of allergy or severe reaction to adhesive or tape that must be used in the study.
8. Use oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, dipeptidyl peptidase-4 (DPP-4) inhibitors, Sodium-glucose Cotransporter-2 (SGLT-2) inhibitors anti-diabetic medications.
9. Any investigational drug use within 30 days prior to enrollment.
10. Pregnant or lactating females.
11. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diva D De Leon, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Arpana Rayannavar, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Russell SJ, El-Khatib FH, Nathan DM, Magyar KL, Jiang J, Damiano ER. Blood glucose control in type 1 diabetes with a bihormonal bionic endocrine pancreas. Diabetes Care. 2012 Nov;35(11):2148-55. doi: 10.2337/dc12-0071. Epub 2012 Aug 24. PMID 22923666
- [Background] El-Khatib FH, Russell SJ, Magyar KL, Sinha M, McKeon K, Nathan DM, Damiano ER. Autonomous and continuous adaptation of a bihormonal bionic pancreas in adults and adolescents with type 1 diabetes. J Clin Endocrinol Metab. 2014 May;99(5):1701-11. doi: 10.1210/jc.2013-4151. Epub 2014 Jan 31. PMID 24483160
- [Background] Russell SJ, Hillard MA, Balliro C, Magyar KL, Selagamsetty R, Sinha M, Grennan K, Mondesir D, Ekhlaspour L, Zheng H, Damiano ER, El-Khatib FH. Day and night glycaemic control with a bionic pancreas versus conventional insulin pump therapy in preadolescent children with type 1 diabetes: a randomised crossover trial. Lancet Diabetes Endocrinol. 2016 Mar;4(3):233-243. doi: 10.1016/S2213-8587(15)00489-1. Epub 2016 Feb 3. PMID 26850709
- [Background] El-Khatib FH, Balliro C, Hillard MA, Magyar KL, Ekhlaspour L, Sinha M, Mondesir D, Esmaeili A, Hartigan C, Thompson MJ, Malkani S, Lock JP, Harlan DM, Clinton P, Frank E, Wilson DM, DeSalvo D, Norlander L, Ly T, Buckingham BA, Diner J, Dezube M, Young LA, Goley A, Kirkman MS, Buse JB, Zheng H, Selagamsetty RR, Damiano ER, Russell SJ. Home use of a bihormonal bionic pancreas versus insulin pump therapy in adults with type 1 diabetes: a multicentre randomised crossover trial. Lancet. 2017 Jan 28;389(10067):369-380. doi: 10.1016/S0140-6736(16)32567-3. Epub 2016 Dec 20. PMID 28007348
- [Background] De Leon DD, Stanley CA. Mechanisms of Disease: advances in diagnosis and treatment of hyperinsulinism in neonates. Nat Clin Pract Endocrinol Metab. 2007 Jan;3(1):57-68. doi: 10.1038/ncpendmet0368. PMID 17179930
- [Derived] Rayannavar A, Mitteer LM, Balliro CA, El-Khatib FH, Lord KL, Hawkes CP, Ballester LS, Damiano ER, Russell SJ, De Leon DD. The Bihormonal Bionic Pancreas Improves Glycemic Control in Individuals With Hyperinsulinism and Postpancreatectomy Diabetes: A Pilot Study. Diabetes Care. 2021 Nov;44(11):2582-2585. doi: 10.2337/dc21-0416. Epub 2021 Sep 13. PMID 34518377
- See also: Children's Hospital of Philadelphia | Congenital Hyperinsulinism Center Website — http://www.chop.edu/centers-programs/congenital-hyperinsulinism-center
- See also: Boston University | Bionic Pancreas Website — http://www.artificialpancreas.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bihormonal Bionic Pancreas Admission | Standard Care Admission
Started (4 days) | 5 (Individuals who were assigned to BHBP admission then SC admission.) | 5 (Individuals who were assigned to SC admission then BHBP admission.)
Washout (Minimum 1 week at home in between study admissions.) | 5 | 5
Completed (4 days) | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequential Admissions: Bihormonal bionic pancreas admission: Four day inpatient admission where participants will have blood sugar managed by the Bihormonal Bionic Pancreas. Blood sugars will be monitored for safety by study staff.
  *before or after* Standard care admission: Four day inpatient admission where participants will have blood sugar managed by the participant's home-glucose control regimen. Blood sugars will be monitored for safety by study staff.
Arm/Group | Sequential Admissions
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 15.1 [7 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Mean Plasma Glucose Level [Mean (Standard Deviation); unit: mmmol/L]
  Bionic Pancreas Admission | 8.3 (0.7)
  Standard Care Admission | 9.0 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Glucose Level.
Description: Mean plasma glucose concentration, as measured by the Continuous glucose monitoring system (CGMS), during the final 2 days of the Bihormonal Bionic Pancreas Admission compared to the Standard Care Admission.
Time Frame: Days 2-3 of each admission
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sequential Admissions
Number analyzed (Participants) | 10
mg/dL
  Bihormonal Bionic Pancreas Admission | 149.666118 (12.7998623)
  Standard Care Admision | 162.574753 (32.2642656)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of screening until the end of the last day of the subject's second admission. This time period ranged from 16 to 38 days, depending on how many days in between admissions they had.
Arm/Group | Bihormonal Bionic Pancreas Admission | Standard Care Admission
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bihormonal Bionic Pancreas Admission (N=5) | Standard Care Admission (N=5)
Intermittent nasuea (Gastrointestinal disorders) | 2 (3) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03303196/Prot_SAP_000.pdf